CLINICAL TRIAL: NCT06905249
Title: Midclavicle Block: A Clinical Observational Study
Acronym: MCB
Status: Completed | Type: Observational
Sponsor: Hospital HM Nou Delfos (Other)
Responsible Party: Principal Investigator, HIPÓLITO LABANDEYRA GONZALEZ, Anesthesiologist, Hospital HM Nou Delfos
Other Study IDs: 25.02.2474-GHM; 25.02.2474-GHM (Registry Identifier: CEIm HM Hospitales)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain Management; Regional Anaesthesia; Ultrasound Guided; Clavicle Fracture
Keywords: Clavicle Fracture; ultrasound guided; Midclavicle Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Midshaft Clavicle Fracture Surgery Cohort: Patients undergoing ultrasound-guided midclavicle block for midshaft clavicle fracture surgery. The study evaluates intraoperative and postoperative pain (VAS), sedation levels (Ramsay), diaphragmatic movement (ultrasound), motor and sensory block of the ipsilateral upper limb, sensory block in the clavicle region, hemodynamic stability (BP, HR, SpO₂), onset time and duration of the block, requirement for rescue analgesia, and the incidence of block-related or systemic complications. Qnox and Qcon indices will be continuously recorded intraoperatively for exploratory purposes. Data collection will cover intraoperative and up to 24-hour postoperative periods.

SUMMARY:
This prospective observational study aims to evaluate the effectiveness and safety of the ultrasound-guided Midclavicle Block (MCB) as an anesthetic and analgesic technique for midshaft clavicle fracture surgery. The primary objective is to assess intraoperative pain control using the Visual Analog Scale (VAS). Secondary outcomes include postoperative pain, sedation levels (Ramsay scale), motor and sensory block of the ipsilateral upper limb, hemidiaphragmatic paralysis, and hemodynamic stability. The requirement for rescue analgesia and the incidence of systemic complications will also be recorded. Intraoperative Qnox and Qcon monitoring will be used to explore potential correlations with pain and sedation levels. Data will be collected intraoperatively and postoperatively for up to 24 hours.

DETAILED DESCRIPTION:
This prospective observational study aims to evaluate the effectiveness of the Midclavicle Block (MCB) as an anesthetic and analgesic technique in patients undergoing clavicle fracture surgery. The primary outcome is intraoperative pain control, assessed using the Visual Analog Scale (VAS) in awake patients, to determine the anesthetic effectiveness of the block.

The MCB will be performed under ultrasound guidance with a linear transducer placed in the sagittal plane immediately posterior to the midclavicle. Local anesthetic will be administered via three injections: two 15 mL injections on either side of the fracture site over the anterosuperior periosteum of the clavicle, and a third 10 mL injection crossing the subclavius muscle toward the posteroinferior region of the periosteum. The total volume of local anesthetic administered will be 40 mL.

Secondary outcomes include:

Postoperative pain, assessed using the VAS at immediate recovery and at 6, 12, and 24 hours postoperatively.

Sedation levels, measured with the Ramsay Sedation Scale at 30 minutes and 2 hours after block placement.

Incidence of hemidiaphragmatic paralysis, evaluated with M-mode ultrasound before and after the block, based on diaphragmatic excursion during deep breathing and sniff testing.

Motor block in the ipsilateral upper limb, scored in five nerve distributions (axillary, musculocutaneous, radial, median, ulnar) at baseline, 30 minutes, and 2 hours post-block.

Sensory block in the ipsilateral upper limb, assessed by pinprick in four dermatomes (C5-C8), scored at 30 minutes and 2 hours.

Sensory block in the clavicular region, evaluated over the sternoclavicular joint, midclavicle, and acromioclavicular joint at 30 minutes and 2 hours.

Requirement for postoperative rescue analgesia within the first 24 hours, including type and dosage.

Continuous intraoperative monitoring of Qnox and Qcon indices, to explore their correlation with nociceptive and sedation levels. Qnox estimates nociceptive response; Qcon estimates level of consciousness.

Incidence of systemic complications related to the block, such as hypotension, bradycardia, nausea, or vomiting.

Block onset time and duration, including the time to perform the MCB and onset of anesthetic effect.

Hemodynamic stability, assessed intraoperatively and up to 2 hours postoperatively, by monitoring non-invasive blood pressure, heart rate, and oxygen saturation. Episodes of hypotension (SBP <90 mmHg or >20% drop from baseline) or bradycardia (HR <50 bpm) will be recorded.

The study will enroll 30 adult patients (ages 18-75) scheduled for clavicle fracture surgery at HM Nou Delfos Hospital. Data collection will span intraoperative and early postoperative periods, up to 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with midshaft clavicle fractures scheduled for surgery.
* ASA I-III.
* Signed informed consent.

Exclusion Criteria:

* Allergy to local anesthetics.
* Coagulopathy or active anticoagulant therapy.
* Infection at the puncture site.
* Pregnant or breastfeeding patients.
* Pre-existing neuromuscular disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with midshaft clavicle fractures undergoing surgery under regional anesthesia at a tertiary-level hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Intraoperative Pain Assessment Using the Visual Analog Scale | Intraoperative period
  Intraoperative pain will be assessed using the Visual Analog Scale (VAS), where 0 indicates no pain and 10 represents the worst imaginable pain. Pain scores will be recorded during the procedure whenever feasible, in awake patients, to evaluate the anesthetic effectiveness of the midclavicle block.

SECONDARY OUTCOMES:
Postoperative Pain Assessment Using Visual Analog Scale | Immediate postoperative period, and at 6, 12, and 24 hours postoperatively
  Postoperative pain will be assessed using the Visual Analog Scale (VAS), which ranges from 0 (no pain) to 10 (worst imaginable pain). Pain scores will be recorded in the immediate postoperative period, as well as at 6, 12, and 24 hours after surgery to evaluate the analgesic efficacy of the midclavicle block throughout the early recovery phase.
Sedation Level Assessed by the Ramsay Sedation Scale | 30 minutes and 2 hours post-block
  Sedation will be assessed at 30 minutes and 2 hours after block performance using the Ramsay Sedation Scale, a widely used clinical tool ranging from 1 (anxious or agitated) to 6 (no response to stimuli). This outcome aims to determine whether patients remain adequately awake and cooperative under regional anesthesia.
Incidence of Hemidiaphragmatic Paralysis Assessed by M-mode Ultrasound | Baseline (pre-block), 30 minutes and 2 hours after the block
  Hemidiaphragmatic function will be evaluated using M-mode ultrasonography before the block and at 30 minutes and 2 hours post-block. The measurement will be performed at the right anterior axillary line in the subcostal area, using the liver as an acoustic window. Diaphragmatic excursion will be measured during deep breathing. Hemidiaphragmatic paralysis is defined as a reduction of more than 50% in diaphragmatic excursion compared to baseline, and/or paradoxical movement during sniff testing.
Assessment of Motor Block in the Ipsilateral Upper Limb | Pre-block (baseline), 30 minutes and 2 hours post-block
  Motor block will be assessed before the block, and at 30 minutes and 2 hours after block performance. The evaluation will include motor function in the distribution of the axillary (shoulder abduction), musculocutaneous (elbow flexion), radial (wrist extension), median (wrist flexion), and ulnar (thumb/finger adduction) nerves. Each nerve will be scored using a 3-point scale:
  0 = normal strength
  1. = paresis
  2. = paralysis
  The total motor block score will range from 0 to 10.
Assessment of Sensory Block in the Ipsilateral Upper Limb | 30 minutes and 2 hours post-block
  Sensory function will be assessed by testing response to pinprick in four dermatomes of the ipsilateral upper limb: C5 (deltoid area), C6 (lateral forearm), C7 (dorsum of the hand), and C8 (medial forearm). A 3-point scale will be used in each area:
  0 = normal sensation
  1. = decreased sensation to pinprick
  2. = no sensation to pinprick Sensory block will be considered effective if a score of 1 or 2 is present in at least two dermatomes.
Assessment of Sensory Block in the Clavicle Region | 30 minutes and 2 hours post-block
  Sensory block will be assessed at 30 minutes and 2 hours after block performance in three anatomical areas: the sternoclavicular joint, midclavicle, and acromioclavicular joint. A 4-point scale will be used:
  0 = no reduction in sensation
  1. = decreased sensitivity to pinprick
  2. = no sensitivity to pinprick
  3. = no tactile sensation
  Sensory block will be considered effective if the score is 2 or 3 in the assessed area.
Requirement for Postoperative Rescue Analgesia. | 24 hours postoperative.
  Assess the need for rescue analgesia within the first 24 postoperative hours, including the type of analgesic administered and the doses required.
Continuous Monitoring of Nociception and Sedation Using Qnox and Qcon | Intraoperative period
  During the surgical procedure, continuous monitoring of the Qnox and Qcon indices will be performed using a neurological state monitor with frontal sensors. The Qnox index provides an objective estimate of the patient's nociceptive response, while the Qcon index estimates the level of consciousness.
Incidence of Intraoperative and Postoperative Systemic Complications Related to the Midclavicle Block | During surgery and up to 24 hours postoperatively.
  The incidence of intraoperative and postoperative systemic complications potentially related to the Midclavicle Block (MCB) will be recorded. These include hypotension, bradycardia, nausea, and vomiting.
Onset Time and Duration of the Midclavicular Block Procedure. | Intraoperative
  Measure the onset time of the midclavicular block after local anesthetic injection, as well as the total time required to perform the technique.
Evaluation of Hemodynamic Stability. | Intraoperative period and up to 2 hours post-block.
  Hemodynamic stability will be assessed intraoperatively and during the immediate postoperative period by monitoring non-invasive blood pressure (NIBP), heart rate (HR), and peripheral oxygen saturation (SpO₂). Any episode of hypotension (defined as a systolic blood pressure <90 mmHg or a decrease of >20% from baseline) or bradycardia (heart rate <50 bpm) will be recorded and treated as per standard protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital HM Nou Delfos, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to institutional policies and ethical considerations.

REFERENCES:
- [Background] Labandeyra H, Valdes-Vilches LF, Prats-Galino A, Sala-Blanch X. Midclavicle block: An anatomical study. Eur J Anaesthesiol. 2025 Feb 1;42(2):122-130. doi: 10.1097/EJA.0000000000002079. Epub 2024 Oct 23. PMID 39444274
- [Background] Heredia-Carques C, Labandeyra H, Castellanos M, Valdes-Vilches LF, Tomas X, Sala-Blanch X. Clavipectoral Fascia and Clavipectoral Fascia Plane Block: To Be or Not to Be. Anesth Analg. 2024 Aug 1;139(2):446-448. doi: 10.1213/ANE.0000000000006837. Epub 2024 Mar 12. No abstract available. PMID 38470823
- [Background] Labandeyra H, Heredia C, Valdes-Vilches LF, Prats-Galino A, Sala-Blanch X. Clavipectoral fascia plane block in midshaft clavicle fractures: A cadaveric study. J Clin Anesth. 2024 Sep;96:111469. doi: 10.1016/j.jclinane.2024.111469. Epub 2024 Apr 27. PMID 38678917
- [Background] Labandeyra H, Heredia-Carques C, Campoy JC, Valdes-Vilches LF, Prats-Galino A, Sala-Blanch X. Clavipectoral fascia plane block spread: an anatomical study. Reg Anesth Pain Med. 2024 May 7;49(5):368-372. doi: 10.1136/rapm-2023-104785. PMID 37699731
- [Background] Labandeyra H, Heredia C, Valdes-Vilches LF, Sala-Blanch X. Clavipectoral Fascia Plane Block: Is This Hyperreality? Anesth Analg. 2022 Oct 1;135(4):e23-e24. doi: 10.1213/ANE.0000000000006150. Epub 2022 Sep 15. No abstract available. PMID 36108196
- [Background] Abu Sabaa MA, Elbadry AA, El Malla DA. Ultrasound-Guided Clavipectoral Block for Postoperative Analgesia of Clavicular Surgery: A Prospective Randomized Trial. Anesth Pain Med. 2022 Mar 8;12(1):e121267. doi: 10.5812/aapm.121267. eCollection 2022 Feb. PMID 35433386
- [Background] Xu G, Su P, Cai B, Liu Y, Jiang D, He Y, Zhou M, Zhang M. Ultrasound-guided superficial cervical plexus block combined with clavipectoral fascial plane block or interscalene brachial plexus block in clavicle surgery: a single-centre, double-blind, randomized controlled trial. J Clin Monit Comput. 2023 Aug;37(4):985-992. doi: 10.1007/s10877-022-00968-1. Epub 2023 Jan 10. PMID 36625982
- [Background] Zhuo Q, Zheng Y, Hu Z, Xiong J, Wu Y, Zheng Y, Wang L. Ultrasound-Guided Clavipectoral Fascial Plane Block With Intermediate Cervical Plexus Block for Midshaft Clavicular Surgery: A Prospective Randomized Controlled Trial. Anesth Analg. 2022 Sep 1;135(3):633-640. doi: 10.1213/ANE.0000000000005911. Epub 2022 Jan 21. PMID 35061634
- [Background] Labandeyra H, Furno JL, Campos JL, Roques Escolar V, Valdes Vilches LF. Ultrasound-guided clavipectoral fascia plane block for middle third clavicular fracture: A case series. Rev Esp Anestesiol Reanim (Engl Ed). 2022 Dec;69(10):683-688. doi: 10.1016/j.redare.2021.12.002. Epub 2022 Nov 4. PMID 36344406
- [Background] Ince I, Kilicaslan A, Roques V, Elsharkawy H, Valdes L. Ultrasound-guided clavipectoral fascial plane block in a patient undergoing clavicular surgery. J Clin Anesth. 2019 Dec;58:125-127. doi: 10.1016/j.jclinane.2019.07.011. Epub 2019 Aug 1. No abstract available. PMID 31377668